CLINICAL TRIAL: NCT07152912
Title: A Comparative Study Between the Impact of Isoflurane and Sevoflurane on Oxidative Stress in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Impact of Isoflurane and Sevoflurane on Oxidative Stress in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman adel ali abd moaty, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD185/2024
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Isoflurane; Sevoflurane; Oxidative Stress; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Iso (Experimental): Patients will receive general anesthesia and maintenance by isoflurane.
  Interventions: Drug: Isoflurane
- Group Sev (Experimental): Patients will receive general anesthesia and maintenance by sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Isoflurane — Patients will receive general anesthesia and maintenance by isoflurane.
  Arms: Group Iso
Drug: Sevoflurane — Patients will receive general anesthesia and maintenance by sevoflurane.
  Arms: Group Sev

SUMMARY:
The primary aim of this work is to assess the impact of exposure to isoflurane or sevoflurane as an inhalation anesthetic on the oxidative stress and inflammatory conditions in patients undergoing elective moderate invasive surgery (laparoscopic cholecystectomy).

DETAILED DESCRIPTION:
Oxidative stress is defined as "an imbalance between oxidants and antioxidants in favour of the oxidants, leading to a disruption of redox signalling and control and/or molecular damage.

Isoflurane, which has been utilized since the 1980s, has a particularly low metabolism rate and solubility, leading to reduced induction of anesthesia during surgery and shortened recovery time after surgery.

Sevoflurane began to be used a decade later and has a lower blood-gas partition coefficient than the other anesthetics, leading to rapid induction of anesthesia and fast awakening after anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical Status I-II.
* Undergoing elective laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* Refusal of participation in the study by patients.
* Diabetes (type I or II), endocrine system, and immune system diseases.
* Chronic infection and sepsis.
* Cardiac condition as classified bythe New York Heart Association (NYHA) > class II.
* Hepatic disease: INR > 1.5, and/or albumin < 2.5 g/dL.
* Renal disease: glomerular filtration rate (GFR) < 85 ml/min.
* Mental and neurological disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum level of superoxide dismutase | 6 months postoperatively
  Serum level of superoxide dismutase (SOD) will be recorded.

SECONDARY OUTCOMES:
Serum level of serum soluble programmed cell death-ligand 1 | 6 months postoperatively
  Serum level of serum soluble programmed cell death-ligand 1 (sPD-L1) will be recorded.
Serum level of nuclear factor erythroid 2-related factor | 6 months postoperatively
  Serum level of nuclear factor erythroid 2-related factor (Nrf2) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.